CLINICAL TRIAL: NCT00023634
Title: An Early Phase Study of an EGFRvIII Peptide Based Vaccine in Patients With EGFRvIII Expressing Cancers
Brief Title: S0114 Vaccine Therapy in Treating Patients With Gastric, Prostate, or Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0114; U10CA032102 (NIH); R01CA082661 (NIH); S0114 (Other: SWOG); UW-106 (Other: University of Washington)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Brain Tumors; Gastric Cancer; Ovarian Cancer; Prostate Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; adenocarcinoma of the prostate; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent adult brain tumor; stage IV prostate cancer; recurrent prostate cancer; adult anaplastic astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Ovarian Epithelial; Astrocytoma | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGFR vaccine with GMCSF (Experimental): EGFR antisense DNA 500 mcg peptide w/GMCSF monthly x 6 m
  Interventions: Biological: GMCSF
- EGFR vaccine with KLH (Experimental): EGFR antisense DNA 500 mcg peptide w/KLH monthly x 6 m
  Interventions: Biological: KLH

INTERVENTIONS:
Biological: KLH — 100 mcg w/EGFRvIII
  Other Names: keyhole limpet
  Arms: EGFR vaccine with KLH
Biological: GMCSF — arm 1: 100 mcg w/EGFRvIII
  Other Names: sargramostim
  Arms: EGFR vaccine with GMCSF

SUMMARY:
RATIONALE: Vaccines made from a peptide may make the body build an immune response to kill cancer cells.

PURPOSE: This phase I trial is studying two different vaccines to treat patients who have gastric, prostate, or ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of EGFRvIII peptide vaccine with sargramostim (GM-CSF) or keyhole limpet hemocyanin (KLH) as adjuvant in patients with EGFRvIII-expressing cancer.
* Determine the preexisting antibody and T-cell responses to EGFRvIII in these patients.
* Determine the antibody and T-cell responses to EGFRvIII peptide after immunization with this vaccine with GM-CSF or KLH as adjuvant.

OUTLINE: Patients are assigned to one of two treatment arms.

* Arm I: Patients receive a vaccine containing EGFRvIII peptide admixed with sargramostim (GM-CSF) intradermally monthly.
* Arm II: Patients receive a vaccine containing EGFRvIII peptide admixed with keyhole limpet hemocyanin subcutaneously monthly.

Treatment in both arms continues for 6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 24 patients (12 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one the following:

  * Stage II-IV gastric cancer
  * Stage IIC-IV ovarian cancer in first complete remission

    * CA 125 normal and stable*
  * Grade III anaplastic astrocytoma
  * Stage IV (M1) prostate adenocarcinoma

    * No small cell variations
    * No biochemical progression after definitive surgery, defined by the following:

      * Prostate-specific antigen more than 0.4 ng/mL which remains elevated on 2 additional measurements at least 2 weeks apart after prostatectomy
      * Three consecutive rises in PSA, each at least 1 month apart after definitive radiotherapy
    * Must be receiving androgen blockade
    * PSA less than 5 ng/mL and stable*
* Documented EGFRvIII expression in primary tumor
* Must have received prior surgery and or chemoradiotherapy for disease (except prostate cancer patients) NOTE: *Stable defined as no increase over 2 measurements at least 28 days apart with the last measurement within the past 28 days

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Performance status:

* Zubrod 0

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* SGOT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* No hepatitis

Renal:

* Not specified

Other:

* No other malignancy in the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* No contraindication to receiving sargramostim (GM-CSF) or KLH-based vaccine products
* No autoimmune disease
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 1 month since prior cytotoxic chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 1 month since prior treatment dose corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered from all prior therapies
* No concurrent enrollment on other phase I studies
* No other concurrent immune modulators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
toxicity | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Montgomery, MD, Study Chair — VA Puget Sound Health Care System
Locations (13):
- United States (13):
  - Bay Regional Medical Center, Bay City, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington